CLINICAL TRIAL: NCT00862017
Title: Effect of Monosodium Glutamate on Gastric Emptying and Postprandial Nitrogen in Healthy Volunteers
Brief Title: Effect of Monosodium Glutamate Supplementation on Gastric Emptying and Postprandial Nitrogen Kinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: AgroParisTech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Basic Science
Other Study IDs: AJI-01
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSG (Experimental): Subjects receive a 6-d supplementation of MSG and are studied on the 7th day in the postprandial period following a standard meal ingestion with 2g MSG
  Interventions: Dietary Supplement: MSg supplementation
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: NaCl supplementation

INTERVENTIONS:
Dietary Supplement: MSg supplementation
  Arms: MSG
Dietary Supplement: NaCl supplementation
  Arms: Control

SUMMARY:
There are receptors to free glutamate in the oral cavity and stomach that may mediate effects of this amino acid on gastrointestinal physiology. The investigators hypothesize that a chronic supplementation of monosodium glutamate (MSG) could modulate gastric emptying and the further metabolism of dietary protein in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI 23 to 28

Exclusion Criteria:

* pregnancy
* allergy to milk protein
* gastrointestinal diseases

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-04

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche sur volontaires, Bobigny, France

REFERENCES:
- [Derived] Boutry C, Matsumoto H, Airinei G, Benamouzig R, Tome D, Blachier F, Bos C. Monosodium glutamate raises antral distension and plasma amino acid after a standard meal in humans. Am J Physiol Gastrointest Liver Physiol. 2011 Jan;300(1):G137-45. doi: 10.1152/ajpgi.00299.2010. Epub 2010 Oct 28. PMID 21030612